CLINICAL TRIAL: NCT03088748
Title: Kinematics in Posterior Cruciate Retaining and Bi-Cruciate Retaining Total Knee Replacements
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: 3187FB WIRB20180745
Record Dates: First submitted 2017-03-16; First posted 2017-03-23 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Arthroplasty, Replacement, Knee; Osteoarthritis, Knee
Keywords: total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Smith & Nephew Journey II PCR TKA: Subjects implanted with a Smith & Nephew Journey II posterior cruciate retaining total knee arthroplasty
  Interventions: Device: Journey II posterior cruciate retaining total knee arthroplasty
- Smith & Nephew Journey II BCR TKA: Subjects implanted with a Smith & Nephew Journey II posterior bi-cruciate retaining total knee arthroplasty
  Interventions: Device: Journey II posterior bi-cruciate retaining total knee arthroplasty

INTERVENTIONS:
Device: Journey II posterior cruciate retaining total knee arthroplasty
  Other Names: Journey II PCR TKA
  Groups: Smith & Nephew Journey II PCR TKA
Device: Journey II posterior bi-cruciate retaining total knee arthroplasty
  Other Names: Journey II BCR TKA
  Groups: Smith & Nephew Journey II BCR TKA

SUMMARY:
The purpose of the study is to acquire kinematic in vivo fluoroscopy data from subjects who were implanted with the Smith & Nephew Journey II posterior cruciate retaining (PCR) total knee arthroplasty (TKA) or Journey II bi-cruciate retaining (BCR) TKA. CMR has previously collected data for the Smith & Nephew BCS TKA and compared these kinematics data to those of normal knees.

DETAILED DESCRIPTION:
The objective for this study is to analyze the in vivo kinematics for subjects implanted with either a Journey II PCR or BCR TKA and compare those patterns to subjects having a normal knee from our previous study and to those patterns from subjects having a Smith & Nephew Journey II BCS TKA.

ELIGIBILITY:
Inclusion Criteria:

* Must have must either a Smith & Nephew Journey II PCR or BCR TKA
* Must be at least three months post-operative
* Must have a Knee Society score of >90 with no ligamentous laxity or pain
* Weigh 250 pounds or less
* Should have good-to-excellent post-operative flexion
* Must be able to perform activities (without aid of any kind) and without pain, walking up and down a ramp, performing a deep knee bend and rising from that kneeling position after the deep knee bend
* Must not have had other surgical procedures conducted within the past six months that will prohibit them from performing the study activities
* Must have body mass index (BMI) of less than 38
* Must be between 40-85 years of age
* Must be willing to sign the Informed Consent (IC) / HIPAA and PHI Release forms to participate in the study

Exclusion Criteria:

* Pregnant, potentially pregnant or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study
* Subjects without the required types of knee implants
* Subjects who are unable to walk up and down a ramp, perform a deep knee bend or rising from that kneeling position without aid or support and without pain
* Subjects who have had other surgical procedures conducted within the past six months that will prohibit them from performing the study activities

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a Smith & Nephew Journey II posterior cruciate retaining (PCR) or a Smith & Nephew Journey II bi-cruciate retaining (BCR) total knee arthroplasty (TKA) implanted by Dr. Harold E. Cates.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Komistek, Principal Investigator — The University of Tennessee
Locations (4):
- United States (4):
  - Erlanger Health System, Chattanooga, Tennessee
  - Tennessee Foundation for Education and Research, Knoxville, Tennessee
  - Tennessee Orthopaedic Clinic, Knoxville, Tennessee
  - The University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Smith & Nephew Journey II PCR TKA: Subjects implanted with a Smith & Nephew Journey II posterior cruciate retaining total knee arthroplasty
  Journey II posterior cruciate retaining total knee arthroplasty
- Smith & Nephew Journey II BCR TKA: Subjects implanted with a Smith & Nephew Journey II posterior bi-cruciate retaining total knee arthroplasty
  Journey II posterior bi-cruciate retaining total knee arthroplasty
Period: Overall Study
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Started | 40 | 10
Completed | 40 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA | Total
Number analyzed (Participants) | 40 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.55) | 62.3 (4.32) | 66.3 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 5 | 32
  Male | 13 | 5 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lateral Kinematics Translations While Ascending Ramp
Description: Anterior Posterior (AP) translations of lateral femoral condyles during activity of walking up a ramp. Data represents the motion of a specific part of the femur bone (in this case lateral femoral condyle) during the specified activity (in this case a ramp up). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
mm | 0.1 (5.9) | -0.4 (3.1)

2. Primary Outcome: Medial Kinematics Translations While Ascending Ramp
Description: Anterior Posterior (AP) translations of medial femoral condyles during activity of walking up a ramp. Data represents the motion of a specific part of the femur bone (in this case medial femoral condyle) during the specified activity (in this case a ramp up). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
mm | -1.8 (3.9) | -2.0 (1.3)

3. Primary Outcome: Axial Rotation While Ascending Ramp
Description: Femorotibial axial rotation during activity of walking up a ramp. Data represents the motion of a specific part of the femur bone (in this case femorotibial axial rotation) during the specified activity (in this case a ramp up). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents external rotation of the femur, and negative represents internal rotation of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
degrees | -2.6 (6.3) | -2.0 (4.0)

4. Primary Outcome: Lateral Kinematics Translations While Descending Ramp
Description: Anterior Posterior (AP) translations of lateral femoral condyles during activity of walking down a ramp. Data represents the motion of a specific part of the femur bone (in this case lateral femoral condyle) during the specified activity (in this case a ramp down). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
mm | 0.1 (6.4) | -6.3 (7.5)

5. Primary Outcome: Medial Kinematics Translations While Descending Ramp
Description: Anterior Posterior (AP) translations of medial femoral condyles during activity of walking down a ramp. Data represents the motion of a specific part of the femur bone (in this case medial femoral condyle) during the specified activity (in this case a ramp down). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
mm | -1.0 (3.4) | -3.2 (3.6)

6. Primary Outcome: Axial Rotation While Descending Ramp
Description: Femorotibial axial rotation during activity of walking down a ramp. Data represents the motion of a specific part of the femur bone (in this case femorotibial axial rotation) during the specified activity (in this case a ramp down). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents external rotation of the femur, and negative represents internal rotation of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
degrees | -1.2 (6.2) | 3.7 (7.1)

7. Primary Outcome: Lateral Kinematics Translations During Deep Knee Bend
Description: Anterior Posterior (AP) translations of lateral femoral condyles during a deep knee bend. Data represents the motion of a specific part of the femur bone (in this case lateral femoral condyle) during the specified activity (in this case a deep knee bend). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
mm | -3.7 (5.8) | -9.4 (6.1)

8. Primary Outcome: Medial Kinematics Translations During Deep Knee Bend
Description: Anterior Posterior (AP) translations of medial femoral condyles during a deep knee bend. Data represents the motion of a specific part of the femur bone (in this case medial femoral condyle) during the specified activity (in this case a deep knee bend). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
mm | 1.0 (4.2) | -4.4 (3.8)

9. Primary Outcome: Axial Rotation During Deep Knee Bend
Description: Femorotibial axial rotation during a deep knee bend. Data represents the motion of a specific part of the femur bone (in this case femorotibial axial rotation) during the specified activity (in this case a deep knee bend). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents external rotation of the femur, and negative represents internal rotation of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
degrees | 5.9 (5.7) | 6.0 (7.0)

10. Primary Outcome: Maximum Flexion During Deep Knee Bend
Description: Maximum weight-bearing femorotibial flexion during a deep knee bend. Data represents the motion of a specific part of the femur bone (in this case femorotibial range of motion) during the specified activity (in this case a deep knee bend). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive values are the only possible values in this case, representing the magnitude of weight-bearing flexion. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
Number analyzed (Participants) | 40 | 10
degrees | 112.3 (14.0) | 105.4 (12.8)

ADVERSE EVENTS:
Time Frame: Baseline. Data is collected only on a single day, and no participant follow-up was collected. Thus, this section describes whether or not there were any adverse events on the single day of data collection
Arm/Group | Smith & Nephew Journey II PCR TKA | Smith & Nephew Journey II BCR TKA
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/10
Other Adverse Events (participants affected / at risk) | 0/40 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT03088748/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT03088748/SAP_001.pdf